CLINICAL TRIAL: NCT03680586
Title: Ultra Low Dose 4 Gy Radiation for Definitive Therapy of Gastric MALT Lymphoma
Brief Title: Ultra Low-Dose Radiation Therapy in Treating Patients With Stage I-IV Stomach MALT Lymphoma
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-0392; NCI-2018-01948 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0392 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2018-09-20; First posted 2018-09-21 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Gastric Mucosa-Associated Lymphoid Tissue Lymphoma
MeSH Terms: interventions — Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (low-dose radiation therapy) (Experimental): Patients undergo low-dose radiation therapy over 2 fractions for 2 consecutive days in the absence of disease progression or unacceptable toxicity. Patients with stable or progressive disease at 12-16 weeks post-treatment, or persistent disease at 1 year may undergo higher-dose radiation therapy at the discretion of treating physician.
  Interventions: Drug: Radiation Therapy

INTERVENTIONS:
Drug: Radiation Therapy — Undergo ultra low-dose radiation
  Other Names: Cancer Radiotherapy; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation

SUMMARY:
This trial studies how well ultra low-dose radiation therapy works in treating patients with stage I-IV stomach mucosa-associated lymphoid tissue (MALT) lymphoma. Ultra low-dose radiation therapy may be able to kill tumor cells and shrink tumors while having fewer side effects in patients with MALT lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the efficacy of ultra-low dose 4 Gy gastric radiation, measured as complete gastric response at one year after 4 Gy treatment in patients with marginal zone lymphoma involving the stomach (mucosa-associated lymphoid tissue [MALT]).

SECONDARY OBJECTIVES:

I. To evaluate distant recurrence of marginal zone lymphoma at one year. II. To evaluate toxicity associated with gastric radiation therapy.

EXPLORATORY OBJECTIVES:

I. To determine if microbiome assessment can predict response to ultra-low dose radiation therapy and evaluate the differences in patient microbiome for patients who respond well and poorly to low dose radiation.

II. To determine if micro-ribonucleic acid (RNA) assessment can predict response to ultra-low dose radiation therapy and evaluate the differences in patient microRNA profiles for patients who respond well and poorly to low dose radiation.

III. To explore the role of magnetic resonance imaging (MRI) for staging gastric MALT lymphoma and for predicting response to ultra-low dose radiation therapy.

IV. To encourage optional co-enrollment on study PA18-0644 to facilitate collection and archiving of blood based biomarkers and microbiome samples for patients receiving ultra low dose radiation therapy.

OUTLINE:

Patients undergo low-dose radiation therapy over 2 fractions for 2 consecutive days in the absence of disease progression or unacceptable toxicity. Patients with stable or progressive disease at 12-16 weeks post-treatment, or persistent disease at 1 year may undergo higher-dose radiation therapy at the discretion of treating physician.

After completion of study treatment, patients are followed up every 3 months for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or older with stage I-IV MALT lymphoma involving the stomach. Other low grade lymphomas including follicular grade I/II and chronic lymphocytic leukemia/small lymphocytic lymphoma (CLL/SLL) are ineligible
* Patients must have biopsy-proven disease within the stomach. Patients with clinical and/or radiographic masses will have dimensions noted prior to therapy
* Patients must have H. pylori testing which is negative within 6 months prior to treatment
* Female patients of childbearing potential must have a negative serum pregnancy test (human chorionic gonadotropin [hCG]) within 2 weeks of protocol entry
* Planned systemic therapy prior to, during, or after gastric radiation therapy is permitted however the timing of systemic therapy will be recorded and patients will be stratified according to receipt of systemic therapy
* Patients must have the ability to give informed consent
* Necessary treatment with antibiotics for reasons unrelated to gastric lymphoma is permitted however the timing and nature of the treatment will be recorded

Exclusion Criteria:

* Patients with aggressive B cell lymphoma histology, including diffuse large B cell lymphoma (DLBCL) and grade 3 follicular lymphoma
* Patients with other histologic subtypes of low grade lymphoma (other than MALT) including chronic lymphocytic leukemia/small lymphocytic lymphoma (CLL/SLL) or follicular lymphoma
* Patients with bulky tumors > 10 cm in any dimension
* Patients with a history of prior radiation to the stomach if re-treatment would exceed known gastric or surrounding critical structure (e.g., bowel, spinal cord) tolerance
* Patients who are pregnant
* Patients with scleroderma are ineligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-02-04 (Actual); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Complete gastric response | Up to 1 year
  The complete response rate at one year will be estimated along with 95% confidence intervals.

SECONDARY OUTCOMES:
Distant recurrence defined as disease progression outside of the stomach that was not present initially | Up to 1 year
  Distant recurrence rate at one year will be estimated along with 95% confidence intervals.
Incidence of acute gastrointestinal toxicity graded according to Common Terminology Criteria for Adverse Events (CTCAE) version (v.) 4.03 | Up to 1 year
  Toxicity data will be summarized by frequency tables.
Incidence of chronic gastrointestinal toxicity graded according to CTCAE v. 4.03 | Up to 1 year
  Toxicity data will be summarized by frequency tables.
Time to local gastric event | Up to 1 year
  Will be estimated using the Kaplan-Meier method.
Time to distant event | Up to 1 year
  Will be estimated using the Kaplan-Meier method.
Tumor response | Up to 1 year
  The tumor responses will be summarized stratified by systemic treatments.

CONTACTS AND LOCATIONS:
Overall Officials: Jillian Gunther, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Gunther JR, Xu J, Bhutani MS, Strati P, Fang PQ, Wu SY, Dabaja BS, Dong W, Bhosale PR, Flowers CR, Nair R, Malpica Castillo L, Fayad L, Iyer SP, Parmer S, Wang M, Lee HJ, Samaniego F, Westin J, Ahmed S, Nze CC, Jain P, Neelapu SS, Rodriguez MA, Chihara D, Nastoupil LJ, Pinnix CC. Response-adapted ultra-low-dose 4 Gy radiation as definitive therapy of gastric MALT lymphoma: a single-centre, pilot trial. Lancet Haematol. 2024 Jul;11(7):e521-e529. doi: 10.1016/S2352-3026(24)00133-9. Epub 2024 Jun 3. PMID 38843856
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org